CLINICAL TRIAL: NCT06033443
Title: The Effect of Collaborative Learning on Students' Creative Thinking Disposition and Self-Regulated Learning in the Nursing Education Course: A Single Group Pre-test Post-test Study
Brief Title: Nursing Education and Collaborative Learning
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Namik Kemal University (Other)
Responsible Party: Principal Investigator, Dilek Erden, Dr., Namik Kemal University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: DERDEN-2
Record Dates: First submitted 2023-09-05; First posted 2023-09-13 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Nursing Education
Keywords: Collaborative Learning; nursing students; creative thinking; self-regulated learning

STUDY DESIGN:
Intervention Model Description: Marmara Creative Thinking Disposition Scale and Self-Regulated Learning Scale for Clinical Nursing Practices will be administered to the students who have been informed about the research, after their individual consent has been obtained. Students participating in the research will take 4 hours of theoretical and 4 hours of clinical practice courses for 12 weeks, and a patient education plan will be created in clinical practices.
Masking Description: The aim of the research was to reduce the bias by using a single-blind technique
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experiment group (Experimental): The experimental group will be given collaborative learning-based nursing education for twelve weeks.
  Interventions: Other: Collaborative Learning Group

INTERVENTIONS:
Other: Collaborative Learning Group — The experimental group is the group that receives nursing education based on collaborative learning.

SUMMARY:
Nursing education; It is the process of gaining cognitive, affective and psychomotor skills. Students gain professional competence by equipping them with these skills. Collaborative learning; It not only increases the interaction between the student and the student, but also allows the student to actively participate in the learning process and take responsibility. Thus, it is expected that the quality of health care services will increase with the graduation of nurses who are equipped in terms of knowledge, professional skills and social skills and who have advanced creativity skills. The aim of the study was to examine the effect of the collaborative learning model-based nursing education course on nursing students' creative thinking tendencies and self-regulated learning skills.

DETAILED DESCRIPTION:
The aim of the study was to examine the effect of the collaborative learning model-based nursing education course on nursing students' creative thinking tendencies and self-regulated learning skills. The research is quasi-experimental with a single-group pretest-posttest design. Hypotheses:

1. Students who receive nursing education with a collaborative learning model have a high disposition to think creatively after education.
2. Students who receive nursing education with a collaborative learning model have high self-regulated learning skills after education.

The universe of the research consisted of 3rd year nursing students studying at a university (N:112). The sample consists of all students who enrolled in the 3rd grade, took the nursing education course, volunteered to participate in the research and attend the course. The training program is based on the collaborative learning model. Students participating in the research will take 4 hours of theoretical and 4 hours of clinical practice courses per week for 12 weeks and a patient education plan will be created in clinical practice. The research will be evaluated with the Marmara Creative Thinking Disposition Scale and the Self-Regulated Learning Scale for Clinical Nursing Practices before the education and after the education

ELIGIBILITY:
Inclusion Criteria:

Third-year students who took the course basics of nursing, internal medicine nursing, physiology, pathology, and who voluntarily participated in the study and were not absent were included in the study.

Exclusion Criteria:

* Students in other classes
* Those who do not volunteer to participate in the research
* Students who are absent

Ages: 19 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 112 (Estimated)
Dates: Start 2023-09-18 (Estimated); Primary Completion 2023-12-08 (Estimated); Study Completion 2023-12-08 (Estimated)

PRIMARY OUTCOMES:
Self-Regulated Learning Scale for Clinical Nursing Practices | 1 week
  The scale developed by Şenol and Orgun (2018); It consists of two sub-dimensions, motivation (seven items), learning strategies (nine items) and 16 questions. The scale is 5-point Likert type ("1: I strongly disagree", "5: I strongly agree"). There is no reverse item in the scale and the minimum score that can be taken from the scale is 16 and the maximum score is 80. The overall reliability of the scale is Cronbach's alpha internal consistency coefficient α = 0.89. As the total score increases, the self-regulated learning of the student increases.

SECONDARY OUTCOMES:
Marmara Creative Thinking Dispositions Scale | 1 week
  The scale developed by Özgenel and Çetin (2017); It consists of six sub-dimensions and 25 questions: self-discipline (five items), novelty seeking (eight items), courage (four items), curiosity (three items), doubt (two items), and flexibility (three items). The scale is 5-point Likert type ("1: Never", "5: Always"). There is no reverse item in the scale and the minimum score that can be taken from the scale is 25 and the maximum score is 125. The overall reliability of the scale is Cronbach's alpha internal consistency coefficient α = 0.87. As the total score increases, the creative thinking dispositions of the student increases.

CONTACTS AND LOCATIONS:
Overall Officials: Dilek Erden, PhD., Principal Investigator — Namik Kemal University

IPD SHARING:
Plan to Share IPD: No